CLINICAL TRIAL: NCT07290036
Title: An Open-label, Randomized, Parallel-group, Noninferiority Study to Evaluate the Pharmacokinetics of Bimekizumab Administered Intravenously or as a Subcutaneous Injection in Participants With Active Psoriatic Arthritis and/or Active Axial Spondyloarthritis
Brief Title: A Study to Learn if Bimekizumab Given in Different Ways is Safe and Moves Similarly Throughout the Body Over Time in Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA0019; 2025-522782-30 (Other: EU CT Number)
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Psoriatic Arthritis; Axial Spondyloarthritis
Keywords: Bimekizumab, BKZ, Phase 1B
MeSH Terms: conditions — Arthritis, Psoriatic; Axial Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab arm 1 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 1 or 2 during the PK Lead-In Phase and dosing regimen 1 or 2 during Treatment Period.
  Interventions: Drug: Bimekizumab regimen 1 iv; Drug: Bimekizumab regimen 2 iv
- Bimekizumab arm 2 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 3 during the PK Lead-In Phase and dosing regimen 3 during Treatment Period.
  Interventions: Drug: Bimekizumab regimen 3 sc

INTERVENTIONS:
Drug: Bimekizumab regimen 1 iv — Participants will receive bimekizumab (BKZ) at pre-specified time points.
  Arms: Bimekizumab arm 1
Drug: Bimekizumab regimen 2 iv — Participants will receive bimekizumab (BKZ) at pre-specified time points.
  Arms: Bimekizumab arm 1
Drug: Bimekizumab regimen 3 sc — Participants will receive bimekizumab (BKZ) at pre-specified time points.
  Arms: Bimekizumab arm 2

SUMMARY:
To demonstrate that bimekizumab administered intravenously is noninferior to subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18+ years old and legally able to consent
2. Have active psoriatic arthritis (PsA) or axial spondyloarthritis (axSpA), suitable for bimekizumab treatment
3. Weigh between 45-100 kg (females) or 50-100 kg (males).
4. Be biologic disease-modifying anti-rheumatic drug (bDMARD)-naïve or have stopped bDMARDs ≥3 months or 5 half-lives ago

Exclusion Criteria:

1. Serious organ system disorders (e.g., heart, liver, kidney, gastrointestinal, neuro)
2. Severe psychiatric issues or substance abuse in the past year
3. Recent or chronic infections, including tuberculosis (TB) or nontuberculous mycobacterium (NTMB)
4. Other inflammatory diseases (e.g., rheumatoid arthritis (RA), lupus, inflammatory bowel disease (IBD))
5. Recent live vaccines (within 8 weeks) or Bacillus Calmette-Guerin (BCG) (within 1 year)
6. Recent use of glucagon-like peptide-1 (GLP-1) agonists (within 28 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2028-04-04 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Steady-state Trough Concentration (Ctrough,ss) at Week 16 | Week 16
  Steady-state trough concentration (Ctrough,ss) will be reported.

SECONDARY OUTCOMES:
Occurrence of treatment-emergent Adverse Events (TEAEs) from Baseline to the end of Safety Follow-Up (SFU) Visit | From Baseline to the end of SFU Visit (up to Week 29)
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A TEAE is defined as any AE with a start on or after the first administration of study intervention and on or before 17 weeks after the final administration of study intervention. This includes AEs that worsen in intensity after the start of study intervention.
Occurrence of treatment-emergent Serious Adverse Events (SAEs) from Baseline to the end of SFU Visit | From Baseline to the end of SFU Visit (up to Week 29)
  An SAE is any untoward medical occurrence that, at any dose, meets 1 or more of the criteria listed: Results in death; Is life-threatening; Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Is a congenital anomaly/birth defect; Other situations: Important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention. A TEAE is defined as any AE with a start on or after the first administration of study intervention and on or before 17 weeks after the final administration of study intervention. This includes AEs that worsen in intensity after the start of study intervention.
Occurrence of TEAEs leading to withdrawal of study intervention | From Baseline to the end of SFU Visit (up to Week 29)
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A TEAE is defined as any AE with a start on or after the first administration of study intervention and on or before 17 weeks after the final administration of study intervention. This includes AEs that worsen in intensity after the start of study intervention. TEAEs leading to withdrawal of IMP of the study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733 (UCB)
Locations (10):
- United States (10):
  - Pa0019 114, Peoria, Arizona
  - Pa0019 127, Apple Valley, California
  - Pa0019 111, Covina, California
  - Pa0019 120, Whittier, California
  - Pa0019 128, Whittier, California
  - Pa0019 113, South Miami, Florida
  - Pa0019 115, Duncansville, Pennsylvania
  - Pa0019 116, Jackson, Tennessee
  - Pa0019 121, Bellevue, Washington
  - Pa0019 130, Beckley, West Virginia

IPD SHARING:
Plan to Share IPD: No
The sponsor does not plan to share IPD.